CLINICAL TRIAL: NCT07183813
Title: Effects of Acupuncture for Anxiety and/or Depression Among Patients With Breast Cancer
Brief Title: Acupuncture for Anxiety/Depression in Patients With Breast Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Yuanjie Sun, Attending physician, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2025-075-KY-01
Record Dates: First submitted 2025-09-14; First posted 2025-09-19 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Anxiety Depression; Breast Cancer; Acupuncture
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electroacupuncture group (Experimental): Acupoints:Bai Hui acupoint, An Mian acupoint, Shang Yin Tang acupoint, Tai Yang acupoint, Tian Shu acupoint, Zu SanLi acupoint, Tai Chong acupoint, Shen Men acupoint.
  Interventions: Device: Electroacupuncture group
- Sham electroacupuncture (SEA) group (Sham Comparator): Acupoints: Bai Hui acupoint, An Mian acupoint, Shang Yin Tang acupoint, Tai Yang acupoint, Tian Shu acupoint, Zu San Li acupoint, Tai Chong acupoint, Shen Men acupoint.
  Interventions: Device: Sham electroacupuncture

INTERVENTIONS:
Device: Electroacupuncture group — The needles will be inserted to 15-40mm in acupoints through adhesive pads. Needles will be lifted, thrusted and twirled gently for 3 times to achieve deqi sensation and manipulated every ten minutes during 30-minute maintenance. The electronic acupuncture apparatus will be connected to the bileteral Taiyang, Anmian and Baihui, with a continuous wave of 2 Hertz (Hz) and an electric current of 1-3 milliampere (mA). Participants receive acupuncture treatment three times a week in the first two weeks and twice a week in the last six weeks.
  Arms: Electroacupuncture group
Device: Sham electroacupuncture — The needle will be inserted to 2-3mm in Bai Hui acupoint. For the remaining acupoints, needles will be inserted into the pad till reaching but without penetrating the skin. Needles will be lifted, thrusted and twirled gently for 3 times to simulate the effects of the needle tip penetrating the skin. The electronic acupuncture apparatus will be connected to the Baihui acupoint, Shang Yin Tang acupoint, and bilateral An Mian acupoints, with a continuous wave of 2 Hertz (Hz) and an electric current of 0.1-0.3 mA. In about 3-5 seconds, the electric current will be turned down. Participants receive acupuncture treatment three times a week in the first two weeks and twice a week in the last six weeks.
  Arms: Sham electroacupuncture (SEA) group

SUMMARY:
The aim of this study is to evaluate the effects and safety of acupuncture on anxiety and/or depression among patients with breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Female, aged 18 to 70 years old;
2. Meeting the diagnostic criteria for breast cancer and at TMN I-III;
3. Having completed specialized active treatment for at least one month;
4. With an ECOG score of 0-2;
5. Mild to moderate anxiety and/or depression;
6. Voluntarily joining this study and signing the informed consent form.

Exclusion Criteria:

1. Starting to take or change the regimen of anti-anxiety and/or -depression disorder medication within one month before enrolment;
2. Received psychological intervention or physical therapy one month before enrolment or planning to use in the next 5 months;
3. With diagnosis of anxiety and/or depression disorder prior to the diagnosis of breast cancer;
4. Patients with suicidal tendencies, bipolar disorder and psychotic symptoms;
5. Patients with severe anxiety and/or depression；
6. Patients received acupuncture treatment within one month before enrolment;
7. Participating in other clinical studies on the treatment of anxiety and/or depression;
8. Combined with severe underlying diseases;
9. Patients with severe skin ulcers;
10. Pregnant or lactating patients;
11. Poor compliance.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
The change from baseline in the total score of Hospital Anxiety and Depression Scale (HADS). | week 8
  The total score of HADS ranges from 0 to 42, with higher scores indicating greater anxiety and depression.

SECONDARY OUTCOMES:
The change from baseline in the total score of HADS. | weeks 4, 12, 16 and 20
  The total score of HADS ranges from 0 to 42, with higher scores indicating greater anxiety and depression.
The change from baseline in the score of HADS-A and HADS-D | weeks 4, 8, 12, 16 and 20
  The HADS score ranges from 0 to 42, with higher scores indicating greater anxiety and depression.
Proportion of participants with a total HADS score less than 15, an HADS-A score of less than or equal to 7, and an HADS-D score of less than or equal to 7 | weeks 4, 8, 12, 16 and 20
  The HADS score ranges from 0 to 42, with higher scores indicating greater anxiety and depression.
Change from baseline in Hamilton Depression Scale-14 | Week 4, 8 and 20
  The Hamilton Depression Scale (HAMD) was developed by Hamilton in 1959 and is a clinical tool used to assess anxiety symptoms. All items use a 5-point rating scale from 0 to 4, with a total score ranging from 0 to 56. The cut-off value is 14 points. Generally, a score of >14 points indicates anxiety, >29 points indicates severe anxiety, and the higher the score, the more severe the anxiety symptoms.
Change from baseline in Hamilton Depression Scale-17 | Week 4, 8 and 20
  The Hamilton Depression Scale (HAMD) was developed by Hamilton in 1960 and is the most commonly used scale in clinical assessment of depressive states. All items are scored on a 5-point scale ranging from 0 to 4. The total score is 68. A score of 8-17 indicates mild depression, 18-24 indicates moderate depression, and a score of ≥25 indicates severe depression.
The change from baseline in the Functional Assessment of Cancer Therapy- General and the Functional Assessment of Cancer Therapy-Breast Cancer (FACT-B) | weeks 4,8 and 20
  The FACT-B is a specific scale designed to measure the quality of life in breast cancer patients. The total score of the questionnaire range from 0 to 144, with higher scores indicating worse quality of life.
The change from baseline in the Fear of Cancer Recurrence Inventory-short form(FCRI-SF) | weeks 4, 8 and 20
  The FCRI-SF score ranges from 0 to 168, with higher scores indicating a higher level of fear of cancer recurrence among cancer patients.
The change from baseline in the brief fatigue inventory (BFI) | weeks 4, 8 and 20
  The BFI score ranges from 0 to 10, with higher scores indicating greater fatigue.
The change from baseline in the Insomnia Severity Index (ISI) | weeks 4, 8 and 20
  The ISI score ranges from 0 to 28, with higher scores indicating Insomnia Severity.
The proportion of responders per the Patient Global Index of Improvement (PGI-I) | weeks 8 and 20
  The PGI-I evaluates the overall treatment effect perceived by patients themselves. The change can be rated in 7 levels, including "very much better", "much better", "a little better", "no change", "a little worse", "much worse" or "very much worse". The score of the scale ranges from 1 to 7.
Collection of cranial MRI images. | baseline and week 8
  Data were acquired at the Department of Radiology using a Magneton Skyra 3.0 T MR scanner.

OTHER OUTCOMES:
Expectance assessment | baseline
  Participants will be asked: How do you expect your anxiety and depression will be in 8 weeks?
Assessment of belief in acupuncture | baseline and week 8
  Participants will be asked the question: Do you think your anxiety and depression may be helped by acupuncture?
Blinding assessment | week 8
  Participants will be asked the question: Do you think you have received traditional electroacupuncture in the past 8 weeks?
Adherence assessment | through study completion, an average of five months
  Adherence will be assessed via counting treatment sessions. Those who complete over 80% treatment sessions will be defined as of good adherence.
Proportion of participants using rescue medicine. | through study completion, an average of five months
  The percentage of patients using other medications or therapies that may affect their anxiety and depression.
Safety assessment | through study completion, an average of five months
  Adverse events and severe adverse events will be recorded in the case report form, whether related to interventions or not.

CONTACTS AND LOCATIONS:
Locations (1):
- Guang'anmen Hospital of China Academy of Chinese Medical Sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
Deidentified participant data and data dictionary will be available with publication until six months after publication.
  Formal request should be sent to puzhisun@163.com with a methodologically sound proposal.
  Researchers whose proposal has been approved will sign a data access agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will be available with publication until until six months after publication.
Access Criteria: Formal request should be sent to puzhisun@163.com with a methodologically sound proposal. Researchers whose proposal has been approved.
  Researchers whose proposal has been approved will sign a data access agreement.